CLINICAL TRIAL: NCT07033520
Title: Effects of Online Mindfulness-Based Cognitive Therapy on Pain, Stress-Related Symptoms, and Functionality in Adults With Chronic Migraine and Adverse Childhood Experiences at the International Hospital of Colombia
Brief Title: Effects of Online Mindfulness Therapy on Pain and Stress in Adults With Chronic Migraine and Adverse Childhood Experiences
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fundación Cardiovascular de Colombia (Other)
Collaborators: Universidad de Santander (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CEI-2025-09350
Record Dates: First submitted 2025-06-13; First posted 2025-06-24 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Chronic Migraine; Adverse Childhood Experiences; Depression; Anxiety; Headache Disorders
Keywords: Mindfulness-Based Cognitive Therapy; MBCT; Trauma; Pain; Headache; Online Psychological Intervention; Migraine; Stress-Related Disorders
MeSH Terms: conditions — Depression; Anxiety Disorders; Headache Disorders; Wounds and Injuries; Pain; Headache; Migraine Disorders

STUDY DESIGN:
Intervention Model Description: This study follows a parallel assignment model with two arms: an intervention group receiving an 8-week online Mindfulness-Based Cognitive Therapy (MBCT) program, and a waitlist control group receiving no intervention during the study period. Participants are randomly assigned to each group and assessed at baseline, post-intervention, and at a 3-month follow-up. The design allows for comparison of outcomes between the two independent groups.
Who Masked: Participant, Care Provider
Masking Description: Participants and their treating neurologists (care providers) are blinded to the allocation group. Group assignment is concealed through coded identifiers, and only the study coordination team has access to the randomization list. All interactions and assessments are conducted without revealing group allocation to ensure unbiased clinical management and participant experience.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness-Based Cognitive Therapy Group (Experimental): Participants in this group will receive an 8-week online Mindfulness-Based Cognitive Therapy (MBCT) intervention. The program includes weekly virtual sessions, guided meditations, and cognitive behavioral strategies aimed at reducing pain and stress-related symptoms in individuals with chronic migraine and adverse childhood experiences.
  Interventions: Behavioral: Online Mindfulness-Based Cognitive Therapy
- Control Group (No Intervention): Participants in this group will not receive any intervention during the study period but will continue with their usual care. After study completion, they will be offered the opportunity to participate in the MBCT program.

INTERVENTIONS:
Behavioral: Online Mindfulness-Based Cognitive Therapy — The intervention consists of an 8-week Online Mindfulness-Based Cognitive Therapy (MBCT) program for adults with chronic migraine and adverse childhood experiences. Participants attend one 90-minute virtual group session per week via video conferencing, led by a trained therapist. Daily home practice is encouraged, including 20-30 minutes of guided mindfulness exercises provided as audio files. The program includes cognitive restructuring, body scans, breathing awareness, and acceptance-based techniques. The intervention is fully remote and requires no in-person contact.
  Other Names: MBCT Online
  Arms: Mindfulness-Based Cognitive Therapy Group

SUMMARY:
This study aims to evaluate the effectiveness of an online Mindfulness-Based Cognitive Therapy (MBCT) program in reducing pain, stress-related symptoms, and improving functionality in adults with chronic migraine and a history of adverse childhood experiences (ACE). Participants will be randomly assigned to either the MBCT intervention group or a control group. The intervention is delivered entirely online over eight weeks. The study hypothesizes that MBCT will result in significant improvements in pain perception and stress-related symptoms compared to the control condition.

DETAILED DESCRIPTION:
This clinical trial investigates the effects of an eight-week Online Mindfulness-Based Cognitive Therapy (MBCT) program on adults diagnosed with chronic migraine who also report a history of adverse childhood experiences (ACEs). The study follows a randomized controlled design with two parallel arms: an intervention group receiving MBCT and a control group on a waitlist. Participants in the MBCT group will engage in weekly online sessions, guided meditation exercises, and cognitive restructuring tasks.

The primary hypothesis is that MBCT will significantly reduce self-reported pain intensity and stress-related symptoms, as well as improve functional impact related to headache, compared to the control group. Assessment tools include validated scales such as the Visual Analog Scale (VAS) for pain, Patient Health Questionnaire-9 (PHQ-9) for depressive symptoms, Generalized Anxiety Disorder 7-item scale (GAD-7), and the Headache Impact Test (HIT-6) to assess headache-related disability and functionality.

Data will be collected at three time points: baseline, post-intervention (8 weeks), and follow-up (3 months after completion). The sample will consist of approximately 60 participants, recruited from the International Hospital of Colombia (IHC) and through digital outreach.

This study is classified as minimal risk and has received ethical approval from the Institutional Review Board (IRB) of Fundación Cardiovascular de Colombia. The intervention is delivered entirely online to ensure accessibility and will not interfere with participants' ongoing neurological treatment plans.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients aged 18 years or older with a diagnosis of chronic migraine according to the International Classification of Headache Disorders (ICHD-3), based on diagnostic criteria updated through 2018.
* Willingness to participate in online sessions from 6:00 PM to 8:00 PM on the scheduled day of the intervention.
* Male and female patients with a score of 4 or higher on the Adverse Childhood Experiences Questionnaire.
* Patients who provide informed consent.

Exclusion Criteria:

* Visual, auditory, cognitive, or functional limitations that prevent understanding of therapeutic activities or the ability to perform home tasks.
* Presence of systemic inflammatory disorders, including rheumatic and autoimmune diseases.
* Active malignancy.
* Pregnancy or breastfeeding at the time of the study.
* Pre-existing neurological conditions (e.g., epilepsy, neuromuscular disorders, metabolic diseases, among others).
* Central nervous system tumors.
* Diagnosis of terminal illnesses that prevent follow-up over time.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2025-10-20 (Estimated); Study Completion 2025-11-20 (Estimated)

PRIMARY OUTCOMES:
Reduction in Pain Intensity Measured by the Visual Analog Scale (VAS) | Baseline, 8 weeks, 3-month follow-up
  Pain intensity will be assessed using a numerical Visual Analog Scale (VAS) ranging from 0 (no pain) to 10 (worst imaginable pain). Participants will self-report their average pain intensity over the past week. The VAS will be administered in digital format at baseline, post-intervention (8 weeks), and 3-month follow-up.

SECONDARY OUTCOMES:
Reduction in Depressive Symptoms Measured by the Patient Health Questionnaire-9 (PHQ-9) | Baseline, 8 weeks, and 3-month follow-up.
  Depressive symptoms will be assessed using the Patient Health Questionnaire-9 (PHQ-9), a validated 9-item self-administered questionnaire. Each item is scored from 0 (not at all) to 3 (nearly every day), yielding a total score from 0 to 27.

OTHER OUTCOMES:
Reduction in Anxiety Symptoms Measured by the Generalized Anxiety Disorder-7 (GAD-7) Scale | Baseline, post-intervention, and 3-month follow-up.
  Anxiety symptoms will be measured using the Generalized Anxiety Disorder 7-item scale (GAD-7), a validated self-report scale. Each item is scored from 0 (not at all) to 3 (nearly every day), with total scores ranging from 0 to 21.
Improvement in Functional Impact of Headache Measured by the Headache Impact Test (HIT-6) | baseline, 8 weeks, and 3-month follow-up.
  The Headache Impact Test (HIT-6) will be used to assess the impact of headache on daily functioning and quality of life. The scale includes 6 items scored on a 5-point Likert scale, yielding a total score between 36 and 78.

CONTACTS AND LOCATIONS:
Overall Officials: Elkin Rene Llanez Anaya, MD, Psychiatrist., Study Director — Universidad de Santander
Locations (1):
- International Hospital of Colombia - Fundación Cardiovascular de Colombia, Bucaramanga, Santander Department, Colombia

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared due to ethical considerations, the minimal-risk nature of the study, and institutional privacy policies.

REFERENCES:
- [Background] Roque-Lopez S, Llanez-Anaya E, Alvarez-Lopez MJ, Everts M, Fernandez D, Davidson RJ, Kaliman P. Mental health benefits of a 1-week intensive multimodal group program for adolescents with multiple adverse childhood experiences. Child Abuse Negl. 2021 Dec;122:105349. doi: 10.1016/j.chiabu.2021.105349. Epub 2021 Oct 7. PMID 34628152
- [Background] Kaliman P, Cosin-Tomas M, Madrid A, Roque Lopez S, Llanez-Anaya E, Papale LA, Alisch RS, Davidson RJ. Epigenetic impact of a 1-week intensive multimodal group program for adolescents with multiple adverse childhood experiences. Sci Rep. 2022 Oct 20;12(1):17177. doi: 10.1038/s41598-022-21246-9. PMID 36266402
- [Background] Webster EM. The Impact of Adverse Childhood Experiences on Health and Development in Young Children. Glob Pediatr Health. 2022 Feb 26;9:2333794X221078708. doi: 10.1177/2333794X221078708. eCollection 2022. PMID 35237713
- [Background] Anto M, Jaffee S, Tietjen G, Mendizabal A, Szperka C. Adverse Childhood Experiences and Frequent Headache by Adolescent Self-Report. Pediatr Neurol. 2021 Aug;121:51-55. doi: 10.1016/j.pediatrneurol.2021.04.004. Epub 2021 Apr 16. PMID 34147819
- [Background] Steiner TJ, Stovner LJ, Birbeck GL. Migraine: the seventh disabler. J Headache Pain. 2013 Jan 10;14(1):1. doi: 10.1186/1129-2377-14-1. No abstract available. PMID 23566305